CLINICAL TRIAL: NCT06635499
Title: A Non-interVentional, multI-center and longiTudinAL Study to Describe the Use of SodIum Zirconium CyclosilicatE (LokelmaTM) in Patients Diagnosed With Hyperkalemia in the Real-world Setting in Spain: VITALIZE Study
Brief Title: VITALIZE.Use and Effectiveness of Sodium Zirconium Cyclosilicate (LokelmaTM) in the Real-world Setting in Spain
Acronym: VITALIZE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9480R00047
Record Dates: First submitted 2024-09-12; First posted 2024-10-10 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Hyperkalaemia
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary Objective(s) & Hypothesis(es)

1. To describe the status of kalaemia in patients treated with SZC in the real-world setting at first visit after treatment initiation.
2. To describe the usual HK management after treatment initiation with SZC in the real-world setting.

Secondary Objective(s) & Hypothesis(es)

1. To describe treatment patterns of patients treated with SZC in the real-world setting, as well as the SZC treatment duration.
2. To describe baseline sociodemographic and clinical characteristics of patients treated with SZC in the real-world setting.
3. To describe the evolution of kalaemia and other clinical parameters as well as mortality in patients treated with SZC in the real-world setting.
4. To describe Healthcare Resource Utilization (HCRU) before and after SZC initiation in patients treated with SZC in the real-world setting.
5. To analyse specific characteristics of use of SZC in the real-world setting according to the medical specialties.

For that purpose, a non-interventional, multicenter, longitudinal study, with secondary data collection has been designed involving 20 Spanish public hospitals ans aiming to include 230 patients (10-12 patients per site) has been designed.

DETAILED DESCRIPTION:
Potassium metabolism disorders are among the most frequent electrolyte disturbances in clinical practice, with a spectrum of variable severity. A normal potassium level is critical for proper muscle, heart, and nerve function. An excessive level of potassium can cause abnormal heart rhythms and interfere with the functioning of skeletal muscles.

Hyperkalaemia is defined by a serum potassium concentration above the upper limit of normal: K+ ≥ 5 or 5.5 mEq/L, according to guidelines. It is considered mild when the potassium concentrations are between 5 to 5.5 mEq/L, moderate between 5.5 and 6 mEq/L, and severe if potassium concentrations are higher than 6 mEq/L. Hyperkalaemia is the most serious electrolyte disturbance because it can cause fatal ventricular arrhythmias in minutes.

In a recent meta-analysis, the pooled prevalence of hyperkalaemia (by any definition/threshold) in all adult patients was 6.3% (95%CI 5.8-6.8%) with an incidence of 2.8 cases per 100 person years, while prevalence and incidence were lower in the general population (1.3% (95%CI 1.0-1.8) and 0.4 per 100 person years, respectively). also found that the prevalence was 7.5% in non-dialysis CKD, 8.3% in diabetes, 8.0% in heart failure and 35% in dialysis-dependent CKD, demonstrating that hyperkalaemia risk is influenced by the presence or absence of underlying comorbid conditions. The incidence of hyperkalaemia also increases in the elderly population treated with drugs that induce hyperkalaemia, such as renin-angiotensin-aldosterone system inhibitors (RAASi): angiotensin-converting enzyme inhibitors (ACEi), angiotensin receptor blockers (ARBs), renin inhibitors, mineralocorticoid receptor antagonists (MRA) or potassium-sparing diuretics.

Sodium Zirconium Cyclosilicate (SZC), commercialized as LokelmaTM, is a potassium binder indicated to treat hyperkalaemia constituted by two treatment phases, an initial correction phase (10 g/3 times daily/oral), which is followed by a maintenance phase once patients reach normokalaemia (after 24-48h) (5g/once daily). LokelmaTM was approved by the European Medicines Agency (EMA) in March 2018 and was launched in Spain in Q2 2021 after having demonstrated its efficacy and safety in different populations, doses, and timelines in several clinical trials.

With the aim of giving greater support to these results and, above all, in the context of the Spanish population, complementary data are needed to understand to what extent the broad group of patients in usual clinical practice achieve normokalaemia and maintain it over the study period after initiation with LokelmaTM. The project's goal is to generate real world evidence about the use and the effectiveness of SZC (LokelmaTM) in Spain, through a retrospective Non- Interventional Study (NIS).

Primary Objective(s) & Hypothesis(es)

1. To describe the status of kalaemia in patients treated with SZC in the real-world setting at first visit after treatment initiation.
2. To describe the usual HK management after treatment initiation with SZC in the real-world setting.

Secondary Objective(s) & Hypothesis(es)

1. To describe treatment patterns of patients treated with SZC in the real-world setting, as well as the SZC treatment duration.
2. To describe baseline sociodemographic and clinical characteristics of patients treated with SZC in the real-world setting.
3. To describe the evolution of kalaemia and other clinical parameters as well as mortality in patients treated with SZC in the real-world setting.
4. To describe Healthcare Resource Utilization (HCRU) before and after SZC initiation in patients treated with SZC in the real-world setting.
5. To analyse specific characteristics of use of SZC in the real-world setting according to the medical specialties.

Exploratory Objective(s) & Hypothesis(es) 1. To describe the characteristics of the SZC responder patient according to potassium levels at first visit.

Safety Objective(s) & Hypothesis(es)

1. To describe adverse events in patients treated with SZC in the real-world setting.

ELIGIBILITY:
Inclusion Criteria:

1. Patient of 18 years of age or older at the time of index date (*).
2. Patient with a diagnosis of hyperkalaemia and/or serum potassium concentration ≥ 5 mmol/L recorded at or before the index date (*).
3. Patients with an estimated glomerular filtration rate (eGFR) less than 45 ml/min/1,73m2 recorded before the index date (*).
4. Patient who has initiated LokelmaTM from May 2021 until 3 months before the start data collection for each site (LokelmaTM must be used on label in accordance with Summary of Product Characteristic (SmPC)).
5. Patient with a baseline measure of serum potassium levels at or within 7 days before the index date (*).
6. Patients with at least one follow-up visit during the study period.
7. Patient with data recorded on electronic health records ≥ 6 month before index date (*).

(*) Index date: Day on which the patient starts treatment with SZC (LokelmaTM).

Exclusion Criteria:

1. Patient presenting pseudohyperkalaemia
2. Patients receiving renal replacement therapy
3. Patient who is pregnant or breastfeeding.
4. Patient who, at the time of inclusion in the study, is participating in a clinical trial that includes the use of K+ binders as an investigational medicinal product (IMP).
5. Patient who has explicitly refused consent to participate in research.
6. Patient medical chart is not available for data extraction or the information in it is not analyzable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study targets enrolment of approximately 230 patients diagnosed with hyperkalaemia who have been treated with LokelmaTM following SmPC from May 2021 up to 3 months before the start of data collection per each site in Spain.
  It is expected to include 20 Spanish public hospitals. Initially, each site will aim to include 10-12 patients; however, the study may turn into competitive if needed to meet the planned timelines.
Sampling Method: Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
To describe the status of kalaemia in patients treated with SZC in the real-world setting at first visit after treatment initiation. | From May 2021 up to 3 months before the start of data collection
To describe the usual HK management after treatment initiation with SZC in the real-world setting. | From May 2021 up to 3 months before the start of data collection

SECONDARY OUTCOMES:
To describe treatment patterns of patients treated with SZC in the real-world setting, as well as the SZC treatment duration. | From May 2021 up to 3 months before the start of data collection
To describe baseline sociodemographic and clinical characteristics of patients treated with SZC in the real-world setting. | From May 2021 up to 3 months before the start of data collection
To describe the evolution of kalaemia and other clinical parameters as well as mortality in patients treated with SZC in the real-world setting. | From May 2021 up to 3 months before the start of data collection
To describe Healthcare Resource Utilization (HCRU) before and after SZC initiation in patients treated with SZC in the real-world setting. | From May 2021 up to 3 months before the start of data collection
To analyze specific characteristics of use of SZC according to the medical specialties | From May 2021 up to 3 months before the start of data collection

OTHER OUTCOMES:
Exploratory Objective: To describe the characteristics of the SZC responder patient according to potassium levels at first visit. | From May 2021 up to 3 months before the start of data collection
Safety Objective: To describe adverse events in patients treated with SZC in the real-world setting. | From May 2021 up to 3 months before the start of data collection

CONTACTS AND LOCATIONS:
Locations (14):
- Spain (14):
  - Research Site, A Coruña
  - Research Site, Asturias
  - Research Site, Badajoz
  - Research Site, Barcelona
  - Research Site, Burgos
  - Research Site, Cadiz
  - Research Site, Córdoba
  - Research Site, Huelva
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Santa Cruz de Tenerife
  - Research Site, Valencia
  - Research Site, Zaragoza

REFERENCES:
- [Result] De Sequera Ortíz P, A. A. (2021). Trastornos del Potasio. Hipopotasemia. En Nefrología al día. S.l (págs. 2659-2606). Lorenzo V., López Gómez JM (Eds).
- [Result] Rose BD, P. T. (2001). Hypokalemia. Clinical physiology of acid-base and electrolyte disorders. New York: McGraw-Hill.
- [Result] Humphrey T, Davids MR, Chothia MY, Pecoits-Filho R, Pollock C, James G. How common is hyperkalaemia? A systematic review and meta-analysis of the prevalence and incidence of hyperkalaemia reported in observational studies. Clin Kidney J. 2021 Dec 2;15(4):727-737. doi: 10.1093/ckj/sfab243. eCollection 2022 Apr. PMID 35371465
- [Result] Larivee NL, Michaud JB, More KM, Wilson JA, Tennankore KK. Hyperkalemia: Prevalence, Predictors and Emerging Treatments. Cardiol Ther. 2023 Mar;12(1):35-63. doi: 10.1007/s40119-022-00289-z. Epub 2022 Dec 12. PMID 36503972
- [Result] Palmer BF, L. M. (1996). Effect of aging on renal function and disease. The Kidney. Philadelphia: Brenner & Rector's.